CLINICAL TRIAL: NCT04821362
Title: Comparison Of Standart Technique, Ultrasonography And Near-Infrared Light In Difficult Peripheral Vascular Access: A Randomised Controlled Trial
Brief Title: Comparison of Different Techniques on First Attempt Success in Difficult Vascular Access Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sercan Yalcinli, Attending Physician, MD, Ege University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18-7/32
Record Dates: First submitted 2019-04-05; First posted 2021-03-29 (Actual); Results first posted 2021-12-03 (Actual); Last update posted 2021-12-03 (Actual); Status verified 2021-10

CONDITIONS: Vascular Access
Keywords: peripheral intravenous catheter; near infrared; ultrasound

STUDY DESIGN:
Intervention Model Description: A prospective, experimental, randomized controlled trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard technique group (No Intervention): In this group, peripheral intravenous catheter insertion will be performed routinely.
- Ultrasound group (Active Comparator): In this group, peripheral intravenous catheter insertion will be performed with ultrasound. A linear probe will be used for procedures.
  Interventions: Device: Ultrasound group
- Near Infrared Device Group (Active Comparator): In this group, peripheral intravenous catheter insertion will be performed with AccuVein AV 400.
  Interventions: Device: Near Infrared Device Group

INTERVENTIONS:
Device: Ultrasound group — In the ultrasound group, the nurses will insert the cannulas to the peripheral veins as horizontally and longitudinally with the linear probe.
  Arms: Ultrasound group
Device: Near Infrared Device Group — In the near infrared device group, the nurses will insert the cannulas to the peripheral veins with AccuVein AV 400.
  Arms: Near Infrared Device Group

SUMMARY:
The aim of this study is to investigate whether there is any difference between the use of standard techniques, ultrasonography and infra-red light for the success of the first attempt in difficult peripheral vascular access patients. Patients who have difficult vascular access history ( often need 2 or more attempt to access peripheral intravenous catheter), who do not have palpable or visible vein after tourniquet, and who have the hard anticipation according to operator ( easy-moderate-hard) are included to study. The primary objective is planned as the determination of the success rate in the first attempt. Secondary aims of the study were determined as: total procedure time,total number of attempts, and need for rescue procedure

DETAILED DESCRIPTION:
Before starting the study, all nurses who work as senior nurse in the emergency department will be informed. All the Emergency Nurses who are willing to participate in the study (the consent form from the nurses who will be included in the study) will be taken pretest to measure their knowledge about ultrasound and infrared light usage for intravenous access. Then, the 4-hours theoretical and 4-hours practical lesson accompanied by an infrared device and a single-operator with horizontal and longitudinal vascular access with ultrasonography will be explained by the experienced Emergency Medicine Specialist to all the senior nurses . Introduction of ultrasonography device in the theoretical training, principles of using, linear probe and its properties, horizontal and longitudinal axis concepts used in the determination of venous structures, principles of determination of venous structures in ultrasonography, differentiation of artery and nerve structures will be explained. The introduction of the device for infrared light, the principles of operation, the distance between the light and operation area and the positioning of the device will be discussed. Practical trainings will be arranged on horizontal and longitudinal axes by using ultrasound on lifeless forearm mannequin. In the practical lesson in the infrared light device, the device will be kept in a proper distance on the live mannequin, being positioned perpendicular to the area to be treated and identification of the vascular structures while the device is operating. After the theoretical and practical training, all of the senior nurses will be evaluated with posttest and the nurses with a success rate of 80% will be included in the study.

Adult patients and/ or their relatives will be included to study if they meet any of the inclusion criteria and accept the consent form. The randomization of the patients according to the number of nurses participating in the study will be determined by the responsible researchers before the study begins. For example, in the study where 10 senior nurses will participate, the number of targeted patients will be at least 270 and 10 boxes specific to each nurse will be created. These boxes will be kept in the senior nurse room. Each box will have 27 different application methods (9 usg, 9 infrared, 9 standard methods). The nurse who accepts to participate in the research will apply the method according to the procedure which will be randomly drawn from this box. In this way, an equal number of procedures will be provided for each nurse and an equal number of procedures will be provided for each nurse.

The application of the procedure on the longitudinal or horizontal axis will be left to senior nurse discretion. In the infrared light approach, 2 applicators will be operated. While holding the auxiliary infra-red light, the practitioner will perform the operation at a distance of 20 cm perpendicular to the process zone. The place of application will be left to the discretion of the practitioner. In order to establish a standard approach between the procedures performed, 18 gauge catheter will be used at the arm and the forearm areas, 20 gauge for the other regions. After the tourniquet is inserted, the procedure time will be calculated as seconds. In order for the successful vascular access to be considered successful, at least 5 ml of blood should be taken or at least 5 ml of saline fluid should be given. In all three approaches, if there is no success after 2 attempts, the 3rd and subsequent trials will be evaluated as rescue interventions and these interventions will be left to the discretion of the practitioner and this will be recorded observably (standard approach, usg, infra red light, central vascular, intraosseous approach, calling senior nurse, calling emergency medicine physician etc.). For all three approaches, the success of the first trial, the total duration of the procedure (in seconds), the total number of trials, and rescue method need will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have previously described a history of difficult vascular access.
* Patients who do not have palpable or visible veins after tourniquet placement or who have been referred to unusual locations due to the lack of appropriate veins in the upper extremity.
* Patients who are expected to be hard to perform the procedure by the senior nurse.

Exclusion Criteria:

* The patients who do not need vascular access.
* Patients who do not give consent
* Pregnant patients
* Patients who are under 18 years old
* Patients who require immediate intervention due to any life-threatening condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Özge Can, MD, Principal Investigator — Ege University; İlhan Uz, MD, Principal Investigator — Ege University; Gülbin Konakçı, Asst. Prof., Principal Investigator — Izmir Demokrasi University
Locations (1):
- Ege University, Izmir, Bornova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keyes LE, Frazee BW, Snoey ER, Simon BC, Christy D. Ultrasound-guided brachial and basilic vein cannulation in emergency department patients with difficult intravenous access. Ann Emerg Med. 1999 Dec;34(6):711-4. doi: 10.1016/s0196-0644(99)70095-8. PMID 10577399
- [Background] Bauman M, Braude D, Crandall C. Ultrasound-guidance vs. standard technique in difficult vascular access patients by ED technicians. Am J Emerg Med. 2009 Feb;27(2):135-40. doi: 10.1016/j.ajem.2008.02.005. PMID 19371518
- [Background] Panebianco NL, Fredette JM, Szyld D, Sagalyn EB, Pines JM, Dean AJ. What you see (sonographically) is what you get: vein and patient characteristics associated with successful ultrasound-guided peripheral intravenous placement in patients with difficult access. Acad Emerg Med. 2009 Dec;16(12):1298-1303. doi: 10.1111/j.1553-2712.2009.00520.x. Epub 2009 Nov 12. PMID 19912132
- [Background] Au AK, Rotte MJ, Grzybowski RJ, Ku BS, Fields JM. Decrease in central venous catheter placement due to use of ultrasound guidance for peripheral intravenous catheters. Am J Emerg Med. 2012 Nov;30(9):1950-4. doi: 10.1016/j.ajem.2012.04.016. Epub 2012 Jul 15. PMID 22795988
- [Background] Parker SI, Benzies KM, Hayden KA, Lang ES. Effectiveness of interventions for adult peripheral intravenous catheterization: A systematic review and meta-analysis of randomized controlled trials. Int Emerg Nurs. 2017 Mar;31:15-21. doi: 10.1016/j.ienj.2016.05.004. Epub 2016 Jul 11. PMID 27411965
- [Background] Aulagnier J, Hoc C, Mathieu E, Dreyfus JF, Fischler M, Le Guen M. Efficacy of AccuVein to facilitate peripheral intravenous placement in adults presenting to an emergency department: a randomized clinical trial. Acad Emerg Med. 2014 Aug;21(8):858-63. doi: 10.1111/acem.12437. PMID 25176152
- [Background] Hanada S, Van Winkle MT, Subramani S, Ueda K. Dynamic ultrasound-guided short-axis needle tip navigation technique vs. landmark technique for difficult saphenous vein access in children: a randomised study. Anaesthesia. 2017 Dec;72(12):1508-1515. doi: 10.1111/anae.14082. Epub 2017 Oct 6. PMID 28983903

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients who need urgent care, <18 years, pregnant, and declined to participate were not included in to study groups.
Period: Overall Study
Arm/Group | Standard Technique Group | Ultrasound Group | Near Infrared Device Group
Started | 90 | 90 | 90
Completed | 90 | 90 | 90
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Technique Group | Ultrasound Group | Near Infrared Device Group | Total
Number analyzed (Participants) | 90 | 90 | 90 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 41 | 49 | 47 | 137
  >=65 years | 49 | 41 | 43 | 133
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68.5 [51 to 76] | 64 [53 to 76] | 64 [49 to 77] | 65 [51 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 51 | 60 | 167
  Male | 34 | 39 | 30 | 103
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 90 | 90 | 90 | 270
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Turkey | 90 | 90 | 90 | 270

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Success in the First Attempt
Description: The success numbers of the first attempt during the implementation of all three methods
Time Frame: From the time of randomization until the time of the first successful attempt, up to 30 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Technique Group | Ultrasound Group | Near Infrared Device Group
Number analyzed (Participants) | 90 | 90 | 90
Participants | 56 | 71 | 53

2. Secondary Outcome: Procedure Time.
Description: Time of the intravenous catheter placement procedure
Time Frame: From the time of the tourniquet application, until the procedure successfully achieved, up to 1 hour.
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | Standard Technique Group | Ultrasound Group | Near Infrared Device Group
Number analyzed (Participants) | 90 | 90 | 90
Seconds | 72 [47 to 134] | 107 [69 to 228] | 82 [61 to 163]

3. Secondary Outcome: Patients Who Need Rescue Methods
Description: The method used as a rescue method when the primary method fails to achieve success.
Time Frame: Up to 1 hour.
Measure: Count of Participants; unit: Participants
Groups:
- Standard Technique Group: The number of patients who need a rescue method in patients who cannot achieve success with the standard method
- Ultrasound Group: The number of patients who need a rescue method in patients who cannot achieve success with the ultrasound method.
- Near Infrared Device Group: The number of patients who need a rescue method in patients who cannot achieve success with the near infrared method
Arm/Group | Standard Technique Group | Ultrasound Group | Near Infrared Device Group
Number analyzed (Participants) | 90 | 90 | 90
Participants | 17 | 17 | 25

4. Secondary Outcome: Number of Attempts
Description: Number of attempts to successfully insert peripheral vascular cateter.
Time Frame: From the time of randomization until the time of the successful attempt, up to 1 hour.
Measure: Median (Inter-Quartile Range); unit: attempts
Arm/Group | Standard Technique Group | Ultrasound Group | Near Infrared Device Group
Number analyzed (Participants) | 90 | 90 | 90
attempts | 1 [1 to 2] | 1 [1 to 1] | 1 [1 to 2]

ADVERSE EVENTS:
Time Frame: 1 hour
Arm/Group | Standard Technique Group | Ultrasound Group | Near Infrared Device Group
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/90 | 0/90
Serious Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/90
Other Adverse Events (participants affected / at risk) | 0/90 | 0/90 | 0/90

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04821362/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04821362/SAP_001.pdf